CLINICAL TRIAL: NCT00575302
Title: Study of Optimal Posology of Gonadotrophins in Patients With Insufficient Ovarian Response Due to Age
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: 36 cases were included and the 4 centers and they are unable to increase their recruitment to obtain the 400 cases necessary to reach statistical significance.
Sponsor: Centre Hospitalier Chretien (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Annick Delvigne, CHC Saint-Vincent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study 300 versus 450
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Infertility
Keywords: IVF; poor responder; recFSH; Fertilization in Vitro; Poor responders
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 300 (Active Comparator): administration of 300 IU Gonal-f® in a short agonist protocol.
  Interventions: Drug: Gonal-f®: follitropin alpha
- 450 (Experimental): administration of 450 IU Gonal-f® in a short agonist protocol.
  Interventions: Drug: Gonal-f®: follitropin alpha

INTERVENTIONS:
Drug: Gonal-f®: follitropin alpha — Gonal-f®: follitropin alpha, administration of 300 U
  Arms: 300
Drug: Gonal-f®: follitropin alpha — Gonal-f®: follitropin alpha, administration of 450 U
  Arms: 450

SUMMARY:
In In vitro fertilization (IVF) treatment, poor responder patients of more than 38 years old are randomized prospectively into two dosages of gonadotrophins. The outcome of treatment will be analyzed.

DETAILED DESCRIPTION:
Women > 38 years, who had an insufficient response to stimulation with regular (for age) posology of 225 IU of gonadotrophins (urinary or recombinant), in an agonist protocol will be randomized prospectively into 2 groups:

300 IU versus 450 IU of Gonal-f® administered in a short agonist protocol. Insufficient response is defined as: development of ≤ 4 mature follicles (of ≥ 16 mm) at time of hCG administration.

Patient can be eligible for several cycles in same protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women > 38 years with insufficient response to stimulation with 225 IU of gonadotrophins (urinary or recombinant), in an agonist protocol.
* Insufficient response is defined as: development of ≤ 4 mature follicles (of ≥ 16 mm) at time of hCG administration.
* Patient can be eligible for several cycles in same protocol.

Exclusion Criteria:

* Patients who already received doses > 225 IU
* Patients older than 42 years
* Patients with basal FSH concentrations ≥ 15 mU/ml at day 3

Ages: 38 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
number of mature oocytes | 1 month

SECONDARY OUTCOMES:
follicular development | 1 month
fertilization rate | 1 month
implantation rate | 1 month
embryo quality | 1 month
pregnancy rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Annick Delvigne, PhD, Principal Investigator — CHC Saint-Vincent
Locations (4):
- Belgium (4):
  - CHC Saint-Vincent, Rocourt, Liège
  - CHU Saint-Pierre, Brussels
  - IMEC, Brussels
  - UZ Gent, Ghent